CLINICAL TRIAL: NCT01845493
Title: Sulforaphane Supplementation in Atopic Asthmatics
Acronym: brasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Michelle Hernandez, MD, Principle Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0056
Record Dates: First submitted 2013-04-17; First posted 2013-05-03 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: asthma; Asthmatics; allergic; allergies
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sulforaphane-rich supplement (Active Comparator): Intervention: broccosprout homogenate (rich in Sulforaphane) taken orally daily x 3 days
  Interventions: Dietary Supplement: Sulforaphane Homogenate
- Alfalfa Sprout Homogenate (Placebo Comparator): Placebo: Alfalfa sprout homogenate taken daily x 3 days (poor in sulforaphane)
  Interventions: Dietary Supplement: Alpha Sprout Homogenate

INTERVENTIONS:
Dietary Supplement: Alpha Sprout Homogenate — Alpha Sprout Homogenate
  Other Names: Placebo
  Arms: Alfalfa Sprout Homogenate
Dietary Supplement: Sulforaphane Homogenate — Active
  Arms: Sulforaphane-rich supplement

SUMMARY:
The investigators will perform a pilot study of daily treatment with oral sulforaphane (SFN) for 3 days to determine if Nuclear factor (erythroid-derived 2)-like 2 (NRF2) induction is possible with this supplementation regimen in individuals with allergic asthma.

DETAILED DESCRIPTION:
This pilot study will examine if oral SFN supplementation can induce NRF2 and NRF2-dependent phase II enzymes in nasal epithelial cells of allergic asthmatics. Subjects will receive both a SFN-rich broccosprout homogenate preparation and an alfalfa sprout homogenate (placebo) in a crossover fashion. mRNA levels of NRF2 and NRF2-dependent phase II enzymes will be compared between the active and placebo periods.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 of both genders
2. History of episodic wheezing, chest tightness, or shortness of breath after age of 6 years consistent with asthma, or physician diagnosed asthma after age of 6 years.
3. AND: Positive methacholine test. A positive test is defined as a provocative concentration of methacholine of 10 mg/ml or less producing a 20% fall in FEV1 (PC20 methacholine). Methacholine challenge in a separate screening protocol (98-0799), or from other venues will be accepted.
4. OR: Pre and post bronchodilator FEV1 improvement by 12% or more after 4 puffs of albuterol inhaler.
5. FEV1 of at least 80% of predicted and FEV1/FVC ratio of at least .70 (without use of bronchodilating medications for 12 hours), consistent with lung function of persons with no more than mild episodic or mild persistent asthma (NHANES III predicted set).
6. Allergic sensitization to at least one of the following allergen preparations: (House Dust Mite f, House dust mite p, Cockroach, Tree mix, Grass Mix, Weed Mix, Mold Mix 1, Mold Mix 2, Rat, Mouse, Guinea Pig, Rabbit, Cat or Dog) confirmed by positive immediate skin test response in a separate screening protocol. Proof of allergy from other venues, including ImmunoCAP testing from a medical workup, provided by the subject, will be accepted.
7. Oxygen saturation of > 94 % and normal blood pressure (Systolic between 150 - 90, Diastolic between 90-60 mm Hg)
8. Willing to provide information regarding health history and habits of cigarette smoke exposure;
9. Willing to avoid antioxidant vitamins and cruciferous vegetables as well as juices/drinks with added vitamin supplements for 2 days prior the baseline screening visit and throughout initial dosing period.
10. Subjects must be willing to avoid antihistamine use for 4 days prior to each session and NSAIDs for 7 days prior to each session. Nasal steroids must be held for 2 weeks prior to the session.

Exclusion Criteria:

1. Medical history or underlying health problems that preclude participation in the protocol per the study physician;
2. Current nutritional disorder such as anorexia, bulimia, irritable bowel syndrome, Crohn's disease etc;
3. Use of oral corticosteroids within the past 4 weeks;
4. Presence of upper or lower respiratory tract infection or treatment with antibiotics within the previous 4 weeks;
5. Pregnancy as determined by menstrual history or urine pregnancy test;
6. Current smokers will be excluded. Anyone with a smoking history > 0.5 pack year and/or >1 pack per month will also be excluded.
7. History of bleeding disorder;
8. Recent nasal surgery (with 6 months). If a subject has had nasal surgery between 6 months and 5 years, a study physician will visualize the area prior to the biopsy to evaluate the suitability of the nose for the procedure.
9. History of intolerance of or aversion to broccoli
10. Unable to withhold nasal steroids for 2 weeks before each session. These subjects may be deferred until after their allergy season.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
mRNA levels of NRF2 and NRF2-dependent phase II enzymes in nasal epithelial cells | 2 hours post third ingestion of SFN/placebo ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Hernandez, MD, Principal Investigator — center for environmental medicine asthma and lung biology
Locations (1):
- Environmental Protection Agency at the University of North Carolina, Chapel Hill, North Carolina, United States